CLINICAL TRIAL: NCT01350830
Title: Early and Late Results of Transinguinal Preperitoneal Patch Repair Versus Anterior Pre-Trasversalis Mesh Repair. A Randomised Study
Brief Title: Preperitoneal Versus Pre-trasversalis Hernia Repair
Acronym: PPTHR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: San Bonifacio Hospital (Other)
Responsible Party: Dept. Surgery, ULSS 20
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHIR-01
Record Dates: First submitted 2011-04-28; First posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-01

CONDITIONS: Direct Inguinal Hernia; Indirect Inguinal Hernia
Keywords: inguinal hernia; groin hernia; chronic pain; mesh repair
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pre-trasversalis mesh repair group (Active Comparator)
  Interventions: Procedure: anterior hernia repair
- trans-inguinal preperitoneal patch group (Active Comparator)
  Interventions: Procedure: transinguinal preperitoneal patch repair

INTERVENTIONS:
Procedure: anterior hernia repair — Inguinal incision is made, external oblique divided and the cord is encircled after identifying ilioinguinal and iliohypogastric nerves. The sac is dissected and reduced, in case of direct hernia the posterior wall of inguinal canal is plicated with polypropylene suture; in presence of indirect hernia the sac is reduced and a stitch is passed in manner that the deep ring is snug about the cord. A pre-shaped mesh is positioned on the floor of the canal around the cord with the two tails overlapping laterally; the mesh is then anchored to the pubic tubercle. External oblique is reapproximated with the cord transposed in the subcutaneous space and skin is sutured.
  Other Names: tension free hernia repair
  Arms: pre-trasversalis mesh repair group
Procedure: transinguinal preperitoneal patch repair — Through a 5-cm inguinal incision external oblique fascia is divided, cremasteric fibers are separated and the elements of the cord are skeletonized. Indirect or direct hernia is approached and through the hernia orifice, the sac is reduced, preperitoneal space is accessed and dissected to allow easily placement of the patch facilitated by the memory recoil ring. In case of indirect hernia the lateral part of patch is split and the two tails sutured around vas and gonadic vessels. Hernia orifice is closed with a polypropylene stitch through transversalis fascia and the mesh; external oblique is closed followed by skin approximation.
  Other Names: Polysoft™ Hernia Patch Bard®
  Arms: trans-inguinal preperitoneal patch group

SUMMARY:
Chronic pain rate is from 0 to 50% after prosthetic groin hernia repair. We compared two anterior technique positioning the mesh in the pre-trasversalis space vs preperitoneal space to assess any differences in term of chronic pain and early and late complications

DETAILED DESCRIPTION:
Chronic pain is evaluated in all presenting types (achy, dull, etc.) moreover foreing body sensation, wall stiffness, paresthesia and numbness are controlled in each patients. Limiting of daily, working, sport and sexual activities (disejaculation) are reported as well.

ELIGIBILITY:
Inclusion Criteria:

* 18 years older

Exclusion Criteria:

* recurrent inguinal hernia
* previous low abdominal operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
chronic pain rate | 6 months
  phone interview and clinic visit

SECONDARY OUTCOMES:
recurrence rate | 2 years
  clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Orcalli, M.D., Study Director — Azienda Ulss 20 Verona
Locations (1):
- San Bonifacio Hospital, San Bonifacio, VR, Italy

REFERENCES:
- [Background] Pelissier EP. Inguinal hernia: preperitoneal placement of a memory-ring patch by anterior approach. Preliminary experience. Hernia. 2006 Jun;10(3):248-52. doi: 10.1007/s10029-006-0079-1. Epub 2006 Apr 21. PMID 16758150
- [Background] Pelissier EP, Monek O, Blum D, Ngo P. The Polysoft patch: prospective evaluation of feasibility, postoperative pain and recovery. Hernia. 2007 Jun;11(3):229-34. doi: 10.1007/s10029-007-0203-x. Epub 2007 Feb 15. PMID 17541701